CLINICAL TRIAL: NCT02026258
Title: Efficiency of Piezotome-Corticision Assisted Orthodontics in Alleviating Mandibular Anterior Crowding - A Randomized Controlled Clinical Trial
Brief Title: Efficiency of Piezotome-Corticision Assisted Orthodontics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Flavio Uribe, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IE-12-047-2
Record Dates: First submitted 2013-12-23; First posted 2014-01-01 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Mandibular Anterior Crowding; Piezocision; Pain Perception
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orthodontics no piezocision (Active Comparator): Subjects will have orthodontic treatment without corticision with piezotome. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-2mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment. The time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Interventions: Device: Orthodontics
- Orthodontics with piezotome corticision (Experimental): Subjects receiving orthodontic treatment in conjunction with piezotome-corticision. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-2mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment. The time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Interventions: Procedure: Piezotome-Corticision; Device: Orthodontics

INTERVENTIONS:
Procedure: Piezotome-Corticision — Local anesthetic will be administered to the labial sulcus of the mandibular incisors. A scalpel will be used to make three vertical incisions through the gingiva, 4mm below the interdental papilla, interproximally between mandibular canines and lateral incisors, and central incisors on the labial aspect of the mandible. The incisions will be 4mm in length. A piezosurgery knife will be used to create the cortical alveolar incisions to a depth of 1mm within the cortical bone. The depth of the cortical incision will be limited to 1mm for a safety margin. Postoperatively, subjects will be advised to rinse with chlorhexidine mouthwash twice a day for one week and take acetaminophen as needed.
  Arms: Orthodontics with piezotome corticision
Device: Orthodontics — Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-2mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment.

SUMMARY:
The aim of this study is to evaluate the hypothesis that a piezotome-corticision procedure will have a transient acceleratory effect on the rate of tooth alignment and the overall treatment time. In addition, the subjects in the piezotome-corticision orthodontics group will experience a different level of pain, comfort, and satisfaction as opposed to the conventional orthodontics group.

DETAILED DESCRIPTION:
This study will specifically try:

1. To compare the time required to achieve complete alignment of crowded mandibular anterior teeth (canine to canine) between piezotome-corticision assisted and conventional orthodontics.
2. To investigate the rate of alignment of mandibular anterior teeth at different time points until complete alignment is achieved using dental casts taken at every visit.
3. To compare subject's perception of pain, comfort and satisfaction between the piezotome-corticision assisted and conventional orthodontics using two questionnaires.

Eligibility criteria includes:

* Adult patients 18 or older
* Single arch or double arch treatment
* Non-extraction treatment in the mandibular arch
* Presence of full complement dentition from first molar to first molar
* No spaces in the mandibular arch
* Mandibular anterior irregularity index greater than 5
* Patient with healthy periodontium and attachment loss of up to 2mm
* The amount of crowding should allow for bracket placement
* No therapeutic intervention planned involving intermaxillary or other intraoral or extraoral appliances including elastics, lip bumpers, maxillary expansion appliances, or headgear prior to the complete alignment of mandibular anterior teeth.

Exclusion criteria includes:

* Failure to provide oral and written consent to participation
* Medical problems that affect tooth movement (Refer to Appendix I)
* Presence of primary teeth in the mandibular anterior area
* Missing permanent mandibular anterior teeth
* Inability to place brackets in the anterior mandibular teeth
* Breakage of any of the mandibular anterior brackets that have not been replaced within a week

Outcome measures

1. Two outcome assessors will be calibrated in the assessment of the Little's irregularity index. The irregularity index will be measured twice by two blinded outcome assessors using a fine-tip digital caliper.
2. The subjects will be instructed to record their level of pain: immediately, 1 hour, 12 hours, and 7 days after the first wire placement [76, 82]. They will be also asked to report if they had taken any pain medications, their level of ease and satisfaction with the procedure, if they would undergo this procedure again, and if they would recommend it to a friend. A 100 mm Visual Analog Scale (VAS) will be used to evaluate the level of pain, ease, and satisfaction of all the subjects, with anchors at each end of the line that read "no pain (easy, satisfied)" (0 mm) and "most pain (complicated, not satisfied)" (100 mm).

ELIGIBILITY:
Inclusion criteria:

* Adult patients 18 or older
* Single arch or double arch treatment
* Non-extraction treatment in the mandibular arch
* Presence of full complement dentition from first molar to first molar
* No spaces in the mandibular arch
* Mandibular anterior irregularity index greater than 5
* Patient with healthy periodontium and attachment loss of up to 2mm
* The amount of crowding should allow for bracket placement
* No therapeutic intervention planned involving intermaxillary or other intraoral or extraoral appliances including elastics, lip bumpers, maxillary expansion appliances, or headgear prior to the complete alignment of mandibular anterior teeth.

Exclusion criteria:

* Failure to provide oral and written consent to participation
* Medical problems that affect tooth movement (Refer to Appendix I)
* Presence of primary teeth in the mandibular anterior area
* Missing permanent mandibular anterior teeth
* Inability to place brackets in the anterior mandibular teeth
* Breakage of any of the mandibular anterior brackets that have not been replaced within a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Uribe, DDS MDS, Principal Investigator — UConn Health
Locations (1):
- Orthodontic Clinic University of Connecticut, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Buschang PH, Campbell PM, Ruso S. Accelerating tooth movement with corticotomies: is it possible and desirable? Semin Orthod 2012;18:286-294.
- [Background] Gameiro GH, Pereira-Neto JS, Magnani MB, Nouer DF. The influence of drugs and systemic factors on orthodontic tooth movement. J Clin Orthod. 2007 Feb;41(2):73-8; quiz 71. No abstract available. PMID 17473406
- [Background] Lee WC. Experimental study of the effect of prostaglandin administration on tooth movement--with particular emphasis on the relationship to the method of PGE1 administration. Am J Orthod Dentofacial Orthop. 1990 Sep;98(3):231-41. doi: 10.1016/s0889-5406(05)81600-2. PMID 2403075
- [Background] Verna C, Dalstra M, Melsen B. The rate and the type of orthodontic tooth movement is influenced by bone turnover in a rat model. Eur J Orthod. 2000 Aug;22(4):343-52. doi: 10.1093/ejo/22.4.343. PMID 11029824
- [Background] Yamasaki K, Shibata Y, Fukuhara T. The effect of prostaglandins on experimental tooth movement in monkeys (Macaca fuscata). J Dent Res. 1982 Dec;61(12):1444-6. doi: 10.1177/00220345820610121401. PMID 6960050
- [Background] Liou EJ, Huang CS. Rapid canine retraction through distraction of the periodontal ligament. Am J Orthod Dentofacial Orthop. 1998 Oct;114(4):372-82. doi: 10.1016/s0889-5406(98)70181-7. PMID 9790320
- [Background] Ren A, Lv T, Kang N, Zhao B, Chen Y, Bai D. Rapid orthodontic tooth movement aided by alveolar surgery in beagles. Am J Orthod Dentofacial Orthop. 2007 Feb;131(2):160.e1-10. doi: 10.1016/j.ajodo.2006.05.029. PMID 17276852
- [Background] Kim SJ, Park YG, Kang SG. Effects of Corticision on paradental remodeling in orthodontic tooth movement. Angle Orthod. 2009 Mar;79(2):284-91. doi: 10.2319/020308-60.1. PMID 19216591
- [Background] Fitzpatrick BN. Corticotomy. Aust Dent J. 1980 Oct;25(5):255-8. doi: 10.1111/j.1834-7819.1980.tb05196.x. PMID 6936001
- [Background] Generson RM, Porter JM, Zell A, Stratigos GT. Combined surgical and orthodontic management of anterior open bite using corticotomy. J Oral Surg. 1978 Mar;36(3):216-9. PMID 272455
- [Background] Gantes B, Rathbun E, Anholm M. Effects on the periodontium following corticotomy-facilitated orthodontics. Case reports. J Periodontol. 1990 Apr;61(4):234-8. doi: 10.1902/jop.1990.61.4.234. PMID 2324923
- [Background] KOLE H. Surgical operations on the alveolar ridge to correct occlusal abnormalities. Oral Surg Oral Med Oral Pathol. 1959 May;12(5):515-29 concl. doi: 10.1016/0030-4220(59)90153-7. No abstract available. PMID 13644913
- [Background] Wilcko WM, Wilcko T, Bouquot JE, Ferguson DJ. Rapid orthodontics with alveolar reshaping: two case reports of decrowding. Int J Periodontics Restorative Dent. 2001 Feb;21(1):9-19. PMID 11829041
- [Background] Chung KR, Kim SH, Lee BS. Speedy surgical-orthodontic treatment with temporary anchorage devices as an alternative to orthognathic surgery. Am J Orthod Dentofacial Orthop. 2009 Jun;135(6):787-98. doi: 10.1016/j.ajodo.2007.03.036. PMID 19524840
- [Background] Frost HM. The regional acceleratory phenomenon: a review. Henry Ford Hosp Med J. 1983;31(1):3-9. No abstract available. PMID 6345475
- [Background] Baloul SS, Gerstenfeld LC, Morgan EF, Carvalho RS, Van Dyke TE, Kantarci A. Mechanism of action and morphologic changes in the alveolar bone in response to selective alveolar decortication-facilitated tooth movement. Am J Orthod Dentofacial Orthop. 2011 Apr;139(4 Suppl):S83-101. doi: 10.1016/j.ajodo.2010.09.026. PMID 21435543
- [Background] Teixeira CC, Khoo E, Tran J, Chartres I, Liu Y, Thant LM, Khabensky I, Gart LP, Cisneros G, Alikhani M. Cytokine expression and accelerated tooth movement. J Dent Res. 2010 Oct;89(10):1135-41. doi: 10.1177/0022034510373764. Epub 2010 Jul 16. PMID 20639508
- [Background] Wang L, Lee W, Lei DL, Liu YP, Yamashita DD, Yen SL. Tisssue responses in corticotomy- and osteotomy-assisted tooth movements in rats: histology and immunostaining. Am J Orthod Dentofacial Orthop. 2009 Dec;136(6):770.e1-11; discussion 770-1. doi: 10.1016/j.ajodo.2009.05.015. PMID 19962598
- [Background] Bogoch E, Gschwend N, Rahn B, Moran E, Perren S. Healing of cancellous bone osteotomy in rabbits--Part I: Regulation of bone volume and the regional acceleratory phenomenon in normal bone. J Orthop Res. 1993 Mar;11(2):285-91. doi: 10.1002/jor.1100110216. PMID 8483041
- [Background] Long H, Pyakurel U, Wang Y, Liao L, Zhou Y, Lai W. Interventions for accelerating orthodontic tooth movement: a systematic review. Angle Orthod. 2013 Jan;83(1):164-71. doi: 10.2319/031512-224.1. Epub 2012 Jun 21. PMID 22720793
- [Background] Wilcko MT, Wilcko WM, Pulver JJ, Bissada NF, Bouquot JE. Accelerated osteogenic orthodontics technique: a 1-stage surgically facilitated rapid orthodontic technique with alveolar augmentation. J Oral Maxillofac Surg. 2009 Oct;67(10):2149-59. doi: 10.1016/j.joms.2009.04.095. PMID 19761908
- [Background] Iino S, Sakoda S, Ito G, Nishimori T, Ikeda T, Miyawaki S. Acceleration of orthodontic tooth movement by alveolar corticotomy in the dog. Am J Orthod Dentofacial Orthop. 2007 Apr;131(4):448.e1-8. doi: 10.1016/j.ajodo.2006.08.014. PMID 17418709
- [Background] Mostafa YA, Mohamed Salah Fayed M, Mehanni S, ElBokle NN, Heider AM. Comparison of corticotomy-facilitated vs standard tooth-movement techniques in dogs with miniscrews as anchor units. Am J Orthod Dentofacial Orthop. 2009 Oct;136(4):570-7. doi: 10.1016/j.ajodo.2007.10.052. PMID 19815161
- [Background] Sanjideh PA, Rossouw PE, Campbell PM, Opperman LA, Buschang PH. Tooth movements in foxhounds after one or two alveolar corticotomies. Eur J Orthod. 2010 Feb;32(1):106-13. doi: 10.1093/ejo/cjp070. Epub 2009 Sep 7. PMID 19736219
- [Background] Cohen G, Campbell PM, Rossouw PE, Buschang PH. Effects of increased surgical trauma on rates of tooth movement and apical root resorption in foxhound dogs. Orthod Craniofac Res. 2010 Aug;13(3):179-90. doi: 10.1111/j.1601-6343.2010.01494.x. PMID 20618720
- [Background] Fischer TJ. Orthodontic treatment acceleration with corticotomy-assisted exposure of palatally impacted canines. Angle Orthod. 2007 May;77(3):417-20. doi: 10.2319/0003-3219(2007)077[0417:OTAWCE]2.0.CO;2. PMID 17465647
- [Background] Aboul-Ela SM, El-Beialy AR, El-Sayed KM, Selim EM, El-Mangoury NH, Mostafa YA. Miniscrew implant-supported maxillary canine retraction with and without corticotomy-facilitated orthodontics. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):252-9. doi: 10.1016/j.ajodo.2009.04.028. PMID 21300255
- [Background] Vercellotti T, Podesta A. Orthodontic microsurgery: a new surgically guided technique for dental movement. Int J Periodontics Restorative Dent. 2007 Aug;27(4):325-31. PMID 17726988
- [Background] Dibart S, Surmenian J, Sebaoun JD, Montesani L. Rapid treatment of Class II malocclusion with piezocision: two case reports. Int J Periodontics Restorative Dent. 2010 Oct;30(5):487-93. PMID 20814602
- [Background] Hernandez-Alfaro F, Guijarro-Martinez R. Endoscopically assisted tunnel approach for minimally invasive corticotomies: a preliminary report. J Periodontol. 2012 May;83(5):574-80. doi: 10.1902/jop.2011.110233. Epub 2011 Sep 26. PMID 21942792
- [Background] Fleming PS, DiBiase AT, Sarri G, Lee RT. Efficiency of mandibular arch alignment with 2 preadjusted edgewise appliances. Am J Orthod Dentofacial Orthop. 2009 May;135(5):597-602. doi: 10.1016/j.ajodo.2007.06.014. PMID 19409342
- [Background] Ngan P, Kess B, Wilson S. Perception of discomfort by patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1989 Jul;96(1):47-53. doi: 10.1016/0889-5406(89)90228-x. PMID 2750720
- [Background] Scheurer PA, Firestone AR, Burgin WB. Perception of pain as a result of orthodontic treatment with fixed appliances. Eur J Orthod. 1996 Aug;18(4):349-57. doi: 10.1093/ejo/18.4.349. PMID 8921656
- [Derived] Uribe F, Davoody L, Mehr R, Jayaratne YSN, Almas K, Sobue T, Allareddy V, Nanda R. Efficiency of piezotome-corticision assisted orthodontics in alleviating mandibular anterior crowding-a randomized clinical trial. Eur J Orthod. 2017 Nov 30;39(6):595-600. doi: 10.1093/ejo/cjw091. PMID 28371882

RESULTS

PARTICIPANT FLOW:
Groups:
- Orthodontics no Piezocision: Subjects will have orthodontic treatment without corticision with piezotome. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-1mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment. The time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Orthodontics: Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-1mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment.
- Orthodontics With Piezotome Corticision: Subjects receiving orthodontic treatment in conjunction with piezotome-corticision. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-1mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment. Time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Piezotome-Corticision: Local anesthetic will be administered to the labial sulcus of the mandibular incisors. A scalpel will be used to make three vertical incisions through the gingiva, 4mm below the interdental papilla, interproximally between mandibular canines and lateral incisors, and central incisors on the labial aspect of the mandible. The incisions will be 4mm in length. A piezosurgery knife will be used to create the cortical alveolar incisions to a depth of 1mm within the cortical bone. The de
Period: Randomized
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision
Started | 20 | 21
Completed | 16 | 19
Not Completed | 4 | 2
Not completed — Did not start treatment | 2 | 1
Not completed — Change in treatment plan | 1 | 0
Not completed — Presence of periodontal disease | 1 | 1
Period: Recieved Allocated Intervention
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision
Started | 16 | 19
Completed | 15 | 17
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Orthodontics no Piezocision: Subjects will have orthodontic treatment without corticision with piezotome. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-2mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment. The time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Orthodontics: Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-1mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment.
- Orthodontics With Piezotome Corticision: Subjects receiving orthodontic treatment in conjunction with piezotome-corticision. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-2mm). The archwire sequence will be the same as the control orthodontic group. The time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Piezotome-Corticision: A piezosurgery knife will be used to create the cortical alveolar incisions to a depth of 1mm within the cortical bone. The depth of the cortical incision will be limited to 1mm for a safety margin.
  Orthodontics: Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-1mm). Archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment.
- Total: Total of all reporting groups
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (9.3) | 30 (12.5) | 29.7 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29
Little Irrgularity at T0 [Mean (Standard Deviation); unit: millimeters] — Little's Irregularity index measures the interproximal contact displacement in mm between the anterior teeth segment from the mesial of the canine on one side to the mesial aspect of the contralateral canine.
  millimeters | 8.32 (2.29) | 6.73 (1.99) | 7.5 (3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days to Complete Alignment of Mandibular Anterior Teeth Based on Little's Irregularity Index
Description: Days until complete alignment of mandibular anterior alignment was achieved after wire insertion on both groups. Complete alignment was based on Little's Irregularity index (Sum of contact displacement in mm between the anterior teeth from mesial of one canine to the mesial of the contralateral canine) of less than 2mm.
Time Frame: From the placement of the first wire to complete alignment of mandibular anteiror teeth, assessed up to 9 months
Measure: Mean (Standard Deviation); unit: Days to complete alignment
Groups:
- Orthodontics no Piezocision: Subjects will have orthodontic treatment without corticision with piezotome. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-1mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment. The time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Orthodontics: Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-2mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment.
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision
Number analyzed (Participants) | 13 | 16
Days to complete alignment | 112 (46.22) | 102.13 (34.73)
Statistical Analysis 1: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; Based on previous findings, it takes approximately 117 ± 46 days for complete alignment of the mandibular anterior teeth in subjects with severe crowding treated without extractions. For a clinically significant 40% faster alignment in the piezotome-corticision group compared to the control group at an alpha-level (p = 0.05) and desired power of 80%, a sample size of 28 subjects (14 per group) was required. Twenty subjects per group assuming an overall attrition rate of 28%; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.52

2. Secondary Outcome: Questionnaires Involving Pain Level
Description: Specific questions questionnaire included:
  1) How much pain/discomfort at the following time points? 1) Immediately after first wire placement (T0), 2) 1 hour, (T1) 3) 12 hrs (T2) and 4) Seven days after (T3). Rated on a scale from 0-100 (No pain-Unbearable pain)
Time Frame: Immediate to 1 week after wire placement (T0-T3)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision
Number analyzed (Participants) | 13 | 16
units on a scale
  Visual Analogue Scale (VAS) at T0 (0-100) | 7.57 (9.65) | 18.25 (24.03)
  VAS T1 | 12.55 (13.67) | 28.74 (25.99)
  VAS T2 | 20.71 (19.09) | 28.93 (18.11)
  VAS T3 | 8.01 (9.06) | 11.46 (14.50)
Statistical Analysis 1: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; VAS T0; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.30
Statistical Analysis 2: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; VAS T1; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.19
Statistical Analysis 3: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; VAS T2; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.19
Statistical Analysis 4: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; VAS T3; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.76

3. Secondary Outcome: Questionnaire on Easiness and Satisfaction With the Procedure
Description: Visual analogue Scale from 0-100
  1. Are you satisfied with your treatment? Very- Not Satisfied (0-100)
  2. How easy was the procedure to you? Easy-Complicated (0-100)
Time Frame: 4-5 weeks after first wire placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision
Number analyzed (Participants) | 13 | 16
units on a scale
  Ease of Procedure | 7.85 (8.79) | 9.35 (10.41)
  Satisfaction with Procedure | 4.31 (8.03) | 9.08 (18.03)
Statistical Analysis 1: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; Ease of Procedure; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.87
Statistical Analysis 2: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; Satisfaction with procedure; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.69

4. Secondary Outcome: Questionnaire Involving Pain Management and Satisfaction With the Procedure
Description: Binomial measurement in questionnaire on medications taken and satisfaction with the procedure
  1. Did you take any pain medication after the procedure? Y/N (Count Yes)
  2. Would you undergo this procedure again? Y/N (Count Yes)
  3. Would you recommend this procedure to a friend? Y/N (Count Yes)
Time Frame: 4-5 weeks after first wire placement
Measure: Count of Participants; unit: Participants
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision
Number analyzed (Participants) | 13 | 16
Participants
  Use of Medications | 8 | 11
  Undergo procedure again | 11 | 14
  Recommend Procedure to Friend | 13 | 14
Statistical Analysis 1: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; Test type: Other; p < 0.05, Fisher Exact; Use of Medications; Fisher chi square = 0.71
Statistical Analysis 2: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; Undergo procedure again; Test type: Other; p < 0.05, Fisher Exact; Fisher chi square = 0.99
Statistical Analysis 3: Comparison: Orthodontics no Piezocision vs Orthodontics With Piezotome Corticision; Recommend procedure to a friend; Test type: Other; p < 0.05, Fisher Exact; Fisher chi square = 0.49

ADVERSE EVENTS:
Time Frame: 3 years, 11 months
Description: Adverse event data collected was based on subjects that had the intervention performed. The number of subjects that received the intervention were 19 for the orthodontics-piezocision group and 16 for the orthodontics- no piezocision group. 0/19 and 0/16 were affected/risk of serious and non-serious adverse events including all-cause mortality. These numbers include drop outs during the trial (3 subjects) and another 3 subjects that were not analyzed in the final analysis.
Groups:
- Orthodontics With Piezotome Corticision: Subjects receiving orthodontic treatment in conjunction with piezotome-corticision. Subjects will be followed every 4-5 weeks after the first wire placement until full alignment of the lower arch (irregularity index 0-2mm). The archwire sequence will be 0.014-in Cu-NiTi wire for the first two visits followed by a 0.014 X 0.025-in Cu-NiTi wire until completion of alignment. The time taken to reach complete alignment for each patient and the rate of tooth alignment will be calculated.
  Piezotome-Corticision: Local anesthetic will be administered to the labial sulcus of the mandibular incisors. A scalpel will be used to make three vertical incisions through the gingiva, 4mm below the interdental papilla, interproximally between mandibular canines and lateral incisors, and central incisors on the labial aspect of the mandible. The incisions will be 4mm in length. A piezosurgery knife will be used to create the cortical alveolar incisions to a depth of 1mm within the cortical bone.
Arm/Group | Orthodontics no Piezocision | Orthodontics With Piezotome Corticision
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

LIMITATIONS AND CAVEATS:
Hi attrition rate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes